CLINICAL TRIAL: NCT03272893
Title: The Effect of Inflammation on Psychological Comorbidity and Behavioral Treatment in Chronic Pain
Brief Title: Biomarkers in Pain and Pain Treatment
Status: Completed | Type: Observational
Sponsor: Rikard Wicksell (Other)
Collaborators: AFA Insurance (Industry); The Swedish Society of Medicine (Other)
Responsible Party: Sponsor-Investigator, Rikard Wicksell, Director of Functional Area Medical Psychology, Karolinska Univ Hospital and head of research group Behavior Medicine, KI, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Other Study IDs: pni-act-2016
Record Dates: First submitted 2017-08-15; First posted 2017-09-06 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Chronic Pain; Inflammation
Keywords: psychoneuroimmunology
MeSH Terms: conditions — Chronic Pain; Inflammation | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The main component in the treatment is exposure to symptoms and feared situations. The iACT program is adapted from the evidence based face-to-face treatment at the Behavioral Medicine unit at Karolinska University Hospital. The iACT program has a different structure but is equal in content to face-to-face treatment, and is to be completed within ten weeks. Participants receive texts, audio files, movies and exercises and have online contact with their psychologist via an internet platform or a smart phone application. The treatment aims to encourage valued behaviors in the presence of inner discomfort.
  Other Names: ACT

SUMMARY:
The goal of this research project is to explore if levels of inflammation predict levels of comorbid mood disorders and treatment success in chronic pain patients. More knowledge in this respect will advance our understanding of chronic pain and comorbid syndromes, and facilitate subgroupings of patients based on the presence and/or level of low-grade inflammation. This research is an important step towards finding an explanation to why treatment effects following behavioral interventions differ across individuals, and generate new hypothesis regarding novel treatment approaches. The specific aims are: 1) to explore if baseline levels of inflammatory biomarkers predict the effects of behavioral intervention and 2) to investigate if baseline levels of inflammatory biomarkers are associated with psychological co-morbidity (e.g. depression, anxiety and fatigue) in patients with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Referred to a specialist clinic within pain management
2. Equal to or older than 18 years
3. Chronic pain (> 6 months)
4. The pain is refractory
5. The pain results in significant functional limitations
6. Stable medication in the last 2 months and no planned changes in medication (except possibly discontinuation or lowering of current dose)

Exclusion Criteria:

1. Spontaneous improvement can be expected (without treatment)
2. Psychiatric comorbidity a) is deemed to be the main reason for the restrictions, or b) should be promptly evaluated and possibly treated, or c) may adversely affect the treatment given in the context of the study
3. Significant risk of suicide
4. Poor teamwork, defined as repeated missed appointments during the assessment / investigation phase
5. Language difficulties (Swedish)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients at the Karolinska Pain Center, suffering from chronic pain that does not respond to any other pain treatments and affects daily functioning severely.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Treatment success | At last psychological session (3 months post baseline)
  The Pain Disability Index

SECONDARY OUTCOMES:
Comorbid psychological problems | At first psychological session (baseline)
  PHQ-9
Blood biomarkers as an effect of treatment | At last psychological session (3 months post baseline)
  Pro-inflammatory cytokines

OTHER OUTCOMES:
Blood biomarkers as predictor for treatment success | At first psychological session (baseline)
  Pro-inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Wicksell, PhD, Principal Investigator — Karolinska Institutet; Bianka Karshikoff, PhD, Study Chair — Karolinska Institutet; Linda Holmström, PhD, Study Chair — Karolinska Institutet; Mats Lekander, PhD, Study Chair — Karolinska Institutet; Jenny Åström, lic psych, Study Chair — Karolinska University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lasselin J, Kemani MK, Kanstrup M, Olsson GL, Axelsson J, Andreasson A, Lekander M, Wicksell RK. Low-grade inflammation may moderate the effect of behavioral treatment for chronic pain in adults. J Behav Med. 2016 Oct;39(5):916-24. doi: 10.1007/s10865-016-9769-z. Epub 2016 Jul 28. PMID 27469518